CLINICAL TRIAL: NCT00360932
Title: An Open-Label Registry Study of the Facial Lipoatrophy Correction Experience With SCULPTRA® in Subjects With Human Immunodeficiency Virus (FACES Study)
Brief Title: Facial Lipoatrophy Correction Experience With SCULPTRA ("FACES" Study)
Acronym: FACES
Status: Completed | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DL6049-0417
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Facial Lipoatrophy
Keywords: facial lipoatrophy; HIV/AIDs
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SCULPTRA (poly-L-lactic acid injection) — Subjects will be treated with SCULPTRA® according to the investigator's judgment, and in accordance with the SCULPTRA® package insert. Details of the exact amount and the time of administration of SCULPTRA® (date, amount, location) will be documented in the CRF at each protocol and non-protocol visit.

SUMMARY:
5 year, open-label study to evaluate safety of SCULPTRA on the signs of lipoatrophy of the face in at least 100 evaluable subjects with human immunodeficiency virus.

ELIGIBILITY:
INCLUSION CRITERIA:

* Subjects seropositive for human immunodeficiency virus;
* In the investigator's judgment, a high probability of 5 year survival and compliance with the study visit schedule;
* Initiating SCULPTRA treatments;
* Ability to comprehend and sign an informed consent document prior to study enrollment.
* No waiver, prospective or retrospective, to deviate in any way from the inclusion/exclusion criteria for clinical study subjects, defined in the study protocol, can be granted to clinical investigators.

EXCLUSION CRITERIA

* Any active skin inflammation or infection in or near the treatment area;
* Any hypersensitivity to the components of SCULPTRA
* Previous treatment with SCULPTRA or any other product for facial lipoatrophy;
* Pregnancy or breastfeeding or anticipating becoming pregnant during the study period; and
* Any other excluding factors that, according to the investigator's judgment, would preclude enrollment in the study.
* No waiver, prospective or retrospective, to deviate in any way from the inclusion/exclusion criteria for clinical study subjects, defined in the study protocol, can be granted to clinical investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects seropositive for human immunodeficiency virus who in the investigator's judgment, have a high probability of 5 year survival and compliance with the study visit schedule, and are initiating SCULPTRA treatments.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2005-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate, by Fitzpatrick skin type and by gender, long-term safety of Poly-L-Lactic acid injection(s) in human immunodeficiency virus subjects with facial lipoatrophy. | 5 years

SECONDARY OUTCOMES:
Evaluate the incidence of hypertrophic scars or keloids in subjects by Fitzpatrick skin types IV-VI, assessed approximately 6 months after completion of treatment; | 5 years
Evaluate the severity, relationship, time to onset, duration, and resolution of adverse events (AEs) by Fitzpatrick skin type and gender; and | 5 years
Evaluate the Quality of Life (QOL) and body image benefit associated with the treatment of facial lipoatrophy. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tara Semanchek, MBA, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States